CLINICAL TRIAL: NCT02578563
Title: SGLT2 Inhibitor Registry in Singapore
Brief Title: Prospective Diabetes Registry of Patients With Type 2 Diabetes Mellitus on SGLT 2 Inhibitor Therapy in Singapore
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1843R00258
Record Dates: First submitted 2015-09-29; First posted 2015-10-19 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate clinical effectiveness and safety of Singaporean Type 2 Diabetes mellitus patients administered SGLT 2 inhibitor monotherapy or in combination with other commonly used hypoglycaemic drugs in real life clinical settings.

To evaluate real life clinical effectiveness and safety of Sodium-Glucose Co-Transporter inhibitor- 2 in Singaporean Type 2 diabetes mellitus patients treated on an outpatient basis in clinical practice setting. The study would also assess treatment patterns with SGLT2 inhibitor patient relevant outcomes in whole population as well as pre identified patient subgroups.

Primary analysis to be done at 1 year and extended analysis at 2 years.

DETAILED DESCRIPTION:
T2DM is associated with overweight/obesity and high fasting plasma glucose (FPG) in White patients, whereas Asian patients are more predisposed to high abdominal fat distribution and high postprandial glucose (PPG) levels, thought to contribute1-4. In response to identical meals, Asian subjects exhibit greater glycemic response than do White subjects4,5. According to the Diabetic Society of Singapore, one out of nine people aged 18 to 69 has diabetes, that's about 11.3% of the population or more than 400,000 people & this is expected to rise with the increasing prevalence of a sedentary lifestyle and high-calorie dietary intake.

SGLT2 inhibitors offers a novel insulin-independent approach to lowering hyperglycaemia and improving metabolic control of type 2 diabetes: they reduce renal glucose reabsorption by inhibition of SGLT2 transporters in the proximal tubule of the kidney, resulting in urinary glucose excretion. Since SGLT2 inhibition is independent of β-cell function or insulin sensitivity, this treatment approach could have applications throughout the natural history of diabetes.6

The reductions in fasting plasma glucose concentration and bodyweight during the treatment with the SGLT2 i, are sustained. Early weight loss, is partly due to a mild osmotic diuresis caused by SGLT2 I, however, the gradual progressive reduction in bodyweight thereafter, with decreased waist circumference, is consistent with a reduction of fat mass. This reduction is potentially attributable to the loss of excess energy through glucose excretion in the urine, an effect supported by the increased urinary glucose/creatinine ratio in patients assigned to SGLT2i.6

Many trials shows that SGLT2 i can improve glycaemic control in patients who have inadequate control with metformin. The drug acts independently of insulin, lowers weight, and is not associated with risk of hypoglycaemia. Safety and tolerability of the drugs were also confirmed. Therefore, addition of SGLT2i to metformin provides a new therapeutic option for treatment of type 2 diabetes.6

Data collection will be done by AZ medical personnel or Pharmacy interns, it will be a paper data collection and will be handed over to the CRO company for data entry & analysis..Data analysis will be done by an independent CRO company namely BioQuest Solutions.

ELIGIBILITY:
Inclusion Criteria:

Patients should meet all of the following criteria at Day 0:

* Outpatient equal to or more than 18 years of age
* Diagnosed as T2DM and treated with antidiabetic medicines at least 3 months and suitable for SGLT2 inhibitor as current treatment judged by PI with HbA1c > 7.0 %
* Will provide completed and signed written informed consents Each participating investigator, will be asked to recruit a fixed number of patients ranging from 10 to 40 depending on site specificities.

Exclusion Criteria:

Patients, with the following criteria will be excluded at Day 0:

* Hypersensitivity to any SGLT2 inhibitor or any of the components in the formulation
* Patients with Type 1 diabetes
* Female patients with gestational diabetes during pregnancy
* Female patients who are pregnant, intending to become pregnant or breastfeeding
* Severe medical condition(s) that in the view of the investigator prohibits participation in the study e.g. cancer, end stage liver disease, end stage renal failure (non-diabetes related)
* Use of other investigational drugs at the time of enrolment
* Renal Function: <30ml/min/1.73m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Simple random sample.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2016-02-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the HbA1c level after 1 year | baseline to 1 year
  to assess whether the therapy initiated with SGLT2 inhibitors at baseline is able to reduce the HbA1c after 1 year.

SECONDARY OUTCOMES:
Change from baseline in FPG level at 6months | Blood samples are collected pre-dose, 6 months post-dose
  By assessment of the other lipid level reduction from baseline lab value to the last lab value
Change from baseline in FPG level at 12months | Blood samples are collected pre-dose, 12 months post-dose
  By assessment of the other lipid level reduction from baseline lab value to the last lab value
Change from baseline in weight at 6months | weight is measured pre-dose, 6 months post-dose
  By assessment of the other weight reduction from baseline value to the last value
Change from baseline in weight at 12 months | weight is measured pre-dose, 12 months post-dose
  By assessment of the other weight reduction from baseline value to the last value
Change from baseline in BP at 6 months | BP is measured pre-dose, 6 months post-dose
  By assessment of the other BP reduction from baseline value to the last value
Change from baseline in BP at 12 months | BP is measured pre-dose, 12 months post-dose
  By assessment of the other BP reduction from baseline value to the last value
Change from baseline in Lipids at 6 months | Blood samples are collected pre-dose, 6 months post-dose
  By assessment of the other lipid level reduction from baseline lab value to the last lab value
Change from baseline in Lipids at 12 months | Blood samples are collected pre-dose, 12 months post-dose
  By assessment of the other lipid level reduction from baseline lab value to the last lab value
Change from baseline in Waist circumference at 6 months | waist circumference is measured pre-dose, 6 months post-dose
  By assessment of the other waist circumference reduction from baseline value to the last value
Change from baseline in Waist circumference at 12 months | waist circumference is measured pre-dose, 12 months post-dose
  By assessment of the other waist circumference reduction from baseline value to the last value

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Singapore, Singapore

REFERENCES:
- [Result] REFERENCES 1. Wang JS, et al. Diabetes Metab Res Rev. 2011;27:79-84 2. Bonora E, et al. Diabetes Care. 2001;24:2023-2029 3. Peter R, et al. Diabet Med. 2006;23:990-995 4. Venn BS, et al. Diabet Med. 2010;27:1205-1208 5. Henry CJ, et al. Br J Nutr. 2008;99:840-845 6. Bailey CJ, et al. Lancet. 2010;375:2223-33
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D1843R00258&attachmentIdentifier=7384e83d-1664-42bf-9058-6140c1ac94e2&fileName=SGLT2i_Study_CSR_28_Dec_2019.pdf&versionIdentifier=